CLINICAL TRIAL: NCT00631605
Title: Studies of Neuroendocrine and Energy Metabolism in Patients With Eating Disorders
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Mei-Chih Tseng/Attending psychiatrist, National Taiwan University Hospital
Other Study IDs: 200705061R
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: eating disorders; ghrelin; leptin; BIA
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This study aims to investigate neuroendocrine, autonomic functioning, and energy metabolism in patients with eating disorder and their relationships with psychopathology of eating disorders (eating patterns, depression, and personality) in these patients.

DETAILED DESCRIPTION:
The study subjects include female patients with DSM-IV diagnosis of AN (n = 30), BN (n = 60) and age-controled normal subjects (n = 30). They will receive a clinical interview and are asked to complete several self-administered questionnaires which included eating-related questionnaires, general psychological functioning scales and personality scales. After overnight fast, each subject undergoes a blood sample collection for neuroendocrine examination, body composition examination using BIA method, basal metabolic rate measurement by indirect calorimetry, and ECG in the morning between 0800 and 0900. Clinical patients would be asked to repeat filling the self-rating scales, weight and body fat measurement, as well as blood drawing again 2 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who fulfilled DSM-IV diagnosis of anorexia nervosa or bulimia nervosa
* Normal controls

Exclusion Criteria:

* Any major psychiatric disorders
* Use of psychoactive medications
* Drug and alcohol abuse
* Medical problems (cardiovascular condition and endocrine disorders)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with eating disorders and normal controls
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2007-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Tseng, MD, Msc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan